CLINICAL TRIAL: NCT03482245
Title: Light Therapy in Patients Undergoing an Operation for a Septic Joint, Necrotizing Soft Tissue Infection, Intraabdominal Sepsis, or Medical Treatment of Pneumonia
Brief Title: The Role of Circadian Clock Proteins in Innate and Adaptive Immunity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Matthew R. Rosengart, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY19030376; 1R01GM145674 (NIH)
Record Dates: First submitted 2018-03-20; First posted 2018-03-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pneumonia; Necrotizing Soft Tissue Infection; Intraabdominal Infections; Infection Joint
Keywords: pneumonia; soft tissue infection; intraabdominal infections; circadian rhythms; blue light; sepsis
MeSH Terms: conditions — Pneumonia; Intraabdominal Infections; Soft Tissue Infections; Sepsis | interventions — Blue Light

STUDY DESIGN:
Intervention Model Description: randomized pilot clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Pneumonia: Blue Light (Experimental): a 12 hours:12 hours light:dark photoperiod cycle of bright (1700 lux) blue (peak 442 nm) enriched light for a total of 3 days after the initial diagnosis and informed consent. The photoperiod is 12 hours: 0800 to 2000. At the transition from light to dark (2000), the blue-enriched light is turned off, and additional blue wavelength light removed with an amber filter.
  Interventions: Other: Blue Light
- Intraabdominal infection: Blue Light (Experimental): a 12 hours:12 hours light:dark photoperiod cycle of bright (1700 lux) blue (peak 442 nm) enriched light for a total of 3 days after the initial diagnosis and informed consent. The photoperiod is 12 hours: 0800 to 2000. At the transition from light to dark (2000), the blue-enriched light is turned off, and additional blue wavelength light removed with an amber filter.
  Interventions: Other: Blue Light
- Necrotizing Soft Tissue Infection: Blue Light (Experimental): a 12 hours:12 hours light:dark photoperiod cycle of bright (1700 lux) blue (peak 442 nm) enriched light for a total of 3 days after the initial diagnosis and informed consent. The photoperiod is 12 hours: 0800 to 2000. At the transition from light to dark (2000), the blue-enriched light is turned off, and additional blue wavelength light removed with an amber filter.
  Interventions: Other: Blue Light
- Pneumonia: Ambient Light (No Intervention): a 12 hours:12 hours light:dark photoperiod cycle of the standard white fluorescent ambient light of the hospital for a total of 3 days after the initial diagnosis and informed consent. The photoperiod is 12 hours: 0800 to 2000. At the transition from light to dark (2000), the ambient white lights are turned off.
- Intraabdominal infection: Ambient Light (No Intervention): a 12 hours:12 hours light:dark photoperiod cycle of the standard white fluorescent ambient light of the hospital for a total of 3 days after the initial diagnosis and informed consent. The photoperiod is 12 hours: 0800 to 2000. At the transition from light to dark (2000), the ambient white lights are turned off.
- Necrotizing Soft Tissue Infection: Ambient Light (No Intervention): a 12 hours:12 hours light:dark photoperiod cycle of the standard white fluorescent ambient light of the hospital for a total of 3 days after the initial diagnosis and informed consent. The photoperiod is 12 hours: 0800 to 2000. At the transition from light to dark (2000), the ambient white lights are turned off.
- Infected Joint: Blue Light (Experimental): a 12 hours:12 hours light:dark photoperiod cycle of bright (1700 lux) blue (peak 442 nm) enriched light for a total of 3 days after the initial diagnosis and informed consent. The photoperiod is 12 hours: 0800 to 2000. At the transition from light to dark (2000), the blue-enriched light is turned off, and additional blue wavelength light removed with an amber filter.
  Interventions: Other: Blue Light
- Infected Joint: Ambient Light (No Intervention): a 12 hours:12 hours light:dark photoperiod cycle of the standard white fluorescent ambient light of the hospital for a total of 3 days after the initial diagnosis and informed consent. The photoperiod is 12 hours: 0800 to 2000. At the transition from light to dark (2000), the ambient white lights are turned off.

INTERVENTIONS:
Other: Blue Light — Subjects that are to be exposed to blue light will be provided by the research personnel with a Day-Light Classic 10,000 lumen SAD light, a device that has been used in many of the previously listed published studies (Epilepsy Behav. 2012 Jul;24(3):359-64. doi: 10.1016/j.yebeh.2012.04.123. Epub 2012 May 30.) The light is small (4 X 16 X 21 inches) and weights less than a pound. It is UV filtered and glare free. There is a single "On/Off" switch. It will be attached to a rolling stand.
  This light is fitted with a blue spectrum filter (peak 442 nm) such that it produces 1700 Lux of blue spectrum lighting when positioned at a distance of 12 inches from the subject. Those subjects assigned to blue light will be asked to shine this small portable blue enriched light on themselves from 0800 to 2000 for 3 days.
  Arms: Infected Joint: Blue Light; Intraabdominal infection: Blue Light; Necrotizing Soft Tissue Infection: Blue Light; Pneumonia: Blue Light

SUMMARY:
Our data suggest that modulating the characteristics of light carries the potential to modify the host response to injury and critical illness and thus, improve outcome. The ability to modify the host response to the stress of major operations and sepsis carries immense potential to improve patient care.

The primary purpose of this study is to determine if exposure to bright blue (442nm) enriched light, by comparison to ambient white fluorescent light, reduces the inflammatory response or organ dysfunction in patients undergoing 1) medical treatment for pneumonia, 2) a 2-stage arthroplasty for surgical management of a septic joint, 3) surgery for a necrotizing soft tissue infection (NSTI), and 4) surgery for an intraabdominal infection (e.g., diverticulitis).

We will expose participants to one of two (2) lighting conditions: 1) high illuminance (~1700 lux,), blue (442nm) spectrum enriched light and 2) ambient white fluorescent light that provides the standard environmental lighting (~300-400 lux, no predominant spectrum) of the hospital.

Both cohorts will be exposed to a 12 hours:12 hours light:dark cycle photoperiod. Those subjects assigned to blue light will be asked to shine this small portable blue enriched light on themselves from 0800 to 2000 for 3 days. At the transition from light to dark, the blue-enriched light is turned off, and additional blue wavelength light removed with an amber filter. Thus, the total period of intervention is 72 hours.

The outcome of interest is change in the inflammatory response after surgery for appendicitis or diverticulitis as measured by the following parameters: white blood cell count, heart rate, the development of abdominal abscess, serum cytokine concentrations.

The outcome of interest is change in the inflammatory response during pneumonia as measured by the following parameters: white blood cell count, heart rate, and serum cytokine concentrations.

DETAILED DESCRIPTION:
The threat of infection is not constant, but rather varies directly with how active we are. This threat is predictable, and for diurnal creatures peaks every 24 hours during the solar day. Not surprising, evolution has prepared us. In the moments preceding daylight, our immune system mobilizes bone marrow leukocytes to populate peripheral tissues and augments leukocyte function. The entire process is orchestrated by the circadian system, and the primary environmental cue is light. Our scientific premise is that the evolutionarily conserved mechanisms of circadian biology confer an immune fitness that can be harnessed and therapeutically applied to treat sepsis.

Within each cell is a circadian clockwork of proteins that dovetails with the molecular machinery regulating cell phenotype. These peripheral clocks are synchronized across the entire organism by the master central clock of the suprachiasmatic nucleus (SCN). Each day, light travels in through the eye to the SCN, and via the autonomic nervous system (ANS), pineal gland, and hypothalamic-pituitary adrenal (HPA) axis, coordinates a temporal program of physiologies, such as enhancing immune competence. This system is maximally entrained by the short wavelength visible blue spectrum. We have applied this blue light in 4 distinct models to reduce tissue injury: ischemia/reperfusion of the liver and kidney, intraabdominal sepsis, and pneumonia. In our studies of sepsis, we identified an optic-parasympathetic pathway through which blue light elevated the expression of the clock protein Rev-Erbalpha within the spleen and bolstered a splenic population of CCR2+ inflammatory monocytes. This enhanced bacterial clearance and increased survival. A Rev-Erbalpha agonist augmented bacterial clearance and prolonged survival, whereas mice deficient in Rev-Erbalpha were no longer protected by blue light, nor were mice that had undergone splenectomy. From these data an innovative paradigm emerges, integrated at the molecular, cellular, and organismal levels, in which circadian pathways regulate cellular clock proteins to optimize the immune niches of the spleen for invading pathogen.

Significance:

Our characterization of the biological mechanisms through which the circadian clock machinery (e.g., Rev-Erbalpha) beneficially alters the cellular response to sepsis provides conceptual and translational innovation to develop novel therapeutics (e.g., blue light) for the treatment of many diseases. It is the logical extension of our prior work showing that blue light in 4 distinct models to reduces enhances immune competence, reduces tissue injury, accelerative bacterial clearance, and improves outcomes: ischemia/reperfusion of the liver and kidney, intraabdominal sepsis, and pneumonia.

Approach:

Subjects will receive the standard preoperative, intraoperative, and postoperative care. All operations will be performed by one of the Trauma/Acute and Critical Care Surgery surgeons at Washington University/Barnes Jewish hospital. Subjects with pneumonia will receive standard medical care for pneumonia. All medical care will be performed by one of the Critical Care Physicians at Washington University/Barnes Jewish hospital. There are no deviations from the standard best practice care received for subjects with these diagnoses.

Discussions of the study, informed consent, and subsequent subject interaction will occur during the initial visit that occurs in the hospital at the time of diagnosis.

Inclusion criteria

Age between 18 and 65 years and one of the following diagnoses:

There are 8 groups that are being evaluation:

1. subjects undergoing an abdominal operation for intraabdominal infection and exposed to Blue light: n=18
2. subjects undergoing an abdominal operation for intraabdominal infection and NOT exposed to Blue light: n=18
3. subjects with pneumonia and exposed to Blue light: n=18
4. subjects with pneumonia and NOT exposed to Blue light: n=18
5. subjects undergoing an operation for a septic joint and exposed to Blue light: n=18
6. subjects undergoing an operation for a septic joint and NOT exposed to Blue light: n=18
7. subjects undergoing an operation for necrotizing soft tissue infection and exposed to Blue light: n=18
8. subjects undergoing an operation for necrotizing soft tissue infection and NOT exposed to Blue light: n=18

Exclusion criteria Subjects who are blind or have sustained traumatic brain injury will not be eligible for participation. The rationale for this exclusion is an inability to determine the integrity of functional optic and suprachiasmatic pathways. Patients who are immunocompromised or immunosuppressed or have been treated for an infection in the prior 30 days will not be eligible for randomization. The rationale for this exclusion is an inability to determine the integrity of the immune response. Patients with an estimated survival of < 48 hours will not be eligible for randomization due to the inability to achieve, and thus assess, the primary outcomes. Patients who test positive for SARS-CoV-2 positive are not eligible, as 1) current standard of care best practices recommend the administration of immunosuppressive medications; and 2) the BSL-2 level classification of our laboratory does not permit us to process biological samples that require this high level of containment.

Intervention We will expose participants to one of two (2) lighting conditions: 1) high illuminance (~1700 lux,), blue (442nm) spectrum enriched light and 2) ambient white fluorescent light that provides the standard environmental lighting (~300-400 lux, no predominant spectrum) of the hospital. The light being used in this study for the intervention of blue light (Day*Light Classic, Uplift Technologies, Dartmouth, NS) is commercially available and is often used to treat such disorders such as seasonal depression and seasonal affective disorder. This device has been used in many of the previously listed published studies (Epilepsy Behav. 2012 Jul;24(3):359-64. doi: 10.1016/j.yebeh.2012.04.123. Epub 2012 May 30.) The light is small, weighs less than a pound, and is portable. It is fitted with a blue filter (Lee filters, Burbank, CA) such that it emits a bright (1700 lux) blue (peak 442 nm spectrum) light at a distance of 12 inches. This intensity of light is 1/5 of what has been used in prior human studies. This illuminance is similar to that of a spring day. Both cohorts will be exposed to a 12 hours:12 hours light:dark cycle photoperiod. Those subjects assigned to blue light will be asked to shine this small portable blue enriched light on themselves from 0800 to 2000 for 3 days. At the transition from light to dark, the blue-enriched light is turned off, and additional blue wavelength light removed with an amber filter. Thus, the total period of intervention is 72 hours. We have used this protocol in a prior IRB-approved and successfully completed study; compliance was 100% with the intervention, and no adverse events were identified.

The comparative groups that are not exposed to Blue light do not receive this light, but otherwise, undergo identical standard of care and will have blood drawn for research purposes.

Group 1: a 12 hours:12 hours light:dark photoperiod cycle of bright (1700 lux) blue (peak 442 nm) enriched light for a total of 3 days after the initial diagnosis (pneumonia) or operation (infected joint, abdominal infection, NSTI).

Group 2: a 12 hours:12 hours light:dark photoperiod cycle of ambient white fluorescent lighting of the hospital for a total of 3 days after the initial diagnosis (pneumonia) or operation (infected joint, abdominal infection, NSTI).

This study is one of effectiveness rather than efficacy. Thus, there are no rigid guidelines that are mandated regarding location or duration of lighting or other environmental restrictions.

Surgical cohort: On the day of surgery, subjects that are to be allocated to Blue light will be exposed to the blue spectrum light after consent and prior to the operation. This light exposure will be initiated, maintained, and removed by the research team. The light will be positioned in front of the subject for the period prior to and for 72 hours during postoperative days 1, 2, and 3 with a 12 hours:12 hours light:dark cycle photoperiod: lights on from 0800 to 2000 for 3 days. At the transition from light to dark, the blue-enriched light is turned off, and additional blue wavelength light removed with an amber filter. At any time the subject may request the light to be removed.

Preoperative and postoperative standard care, including blood sample analysis will be directed by the surgical team and performed at Washington University/Barnes Jewish hospital.

Pneumonia cohort: On the day of diagnosis of pneumonia, subjects that are to be allocated to Blue light will be exposed to the blue spectrum light after consent and prior to the operation. This light exposure will be initiated, maintained, and removed by the research team. The light will be positioned in front of the subject for the period prior to and for 72 hours during postoperative days 1, 2, and 3 with a 12 hours:12 hours light:dark cycle photoperiod: lights on from 0800 to 2000 for 3 days. At the transition from light to dark, the blue-enriched light is turned off, and additional blue wavelength light removed with an amber filter. At any time the subject may request the light to be removed.

For ALL subjects we will abstract laboratory data from the electronic health record.

Six (6) small (1/2 teaspoon) samples of blood will be obtained for research purposes only to measure serum cytokine concentrations. These blood samples are obtained from ALL subjects in the study over the 3 days.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age and less than or equal to 65 years of age
* one of the following diagnoses requiring inpatient hospital care

  1. an operation for intraabdominal infection
  2. an operation for necrotizing soft tissue infection
  3. an operation for an infected joint
  4. medical treatment of pneumonia.

Exclusion Criteria:

* traumatic brain injury
* blindness
* immunocompromised or immunosuppressed state
* infection requiring treatment in preceding 30 days
* blindness
* SARS-CoV-2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pneumonia: change in bronchoalveolar lavage (BAL) bacteria concentration | comparing time of randomization and at 72 hours after randomization
  quantification of the change in bacterial colony forming units (CFU) in BAL fluid
All groups: change in expression of circadian proteins in circulating immune cells | comparing time of randomization and at 72 hours after randomization
  quantification of the change in blood white blood cell counts
All Cohorts: change in serum concentrations of circulating inflammatory mediators in the blood | comparing time of randomization and at 72 hours after randomization
  quantification of change in serum cytokine concentrations

SECONDARY OUTCOMES:
Pneumonia: need for and duration of mechanical ventilation | comparing time of randomization to 28 days
  quantification of days on the ventilator
All Cohorts: change in organ dysfunction | comparing time of randomization and at 72 hours after randomization
  quantification of change in organ dysfunction using the Sequential Organ Failure Assessment scale
Appendicitis and Diverticulitis: intraabdominal abscess formation | from time of randomization to 28-days after randomization
  rate of development of intraabdominal abscess as measured by #subjects/total subjects

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Rosengart, MD MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States